CLINICAL TRIAL: NCT04483648
Title: Effect of Cervical Stabilization Exercises on Cervical Position Error in Patients With Spondyloarthritis: A Randomized Controlled Trial
Brief Title: Cervical Stabilization Exercises in Patients With Spondyloarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Deniz Bayraktar, Assistant Professor, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SpAJPE
Record Dates: First submitted 2020-07-21; First posted 2020-07-23 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Spondyloarthritis
Keywords: Arthritis; Exercise; Proprioception
MeSH Terms: conditions — Spondylarthritis; Arthritis; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Experimental): A progressive home-based cervical stabilization exercise program was delivered by sending messages and video instructions via a freeware and cross-platform messaging service (WhatsApp Messenger) in a weekly basis.
  Interventions: Other: Exercise
- Control Group (No Intervention): Patients in control group did not receive any exercise intervention.

INTERVENTIONS:
Other: Exercise — Home exercises were performed three times in a week for six weeks. Home exercises included range of motion exercises, coordination exercises and strengthening exercises. Repeats and durations of the exercises increased every week to provide progression.
  Arms: Exercise Group

SUMMARY:
The aim of this study is to investigate the effectiveness of cervical stabilization exercises on cervical positioning error in spondyloarthritis patients.

DETAILED DESCRIPTION:
The position sense and kinesthesia are defined as proprioception. In other words, proprioception allows being aware of positions of the body parts in the space. Muscles, tendons, joint capsules are source of proprioception.

Possible damage to these structures due to inflammation may cause diminished proprioception sense. Decreased proprioception was shown for cervical region in axial spondyloarthritis patients in a recent study.

Different exercise programs may help increasing proprioception. Therefore, the aim of the present study is investigate the effects of cervical stabilization exercises on cervical proprioception accuracy.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed as axial spondyloarthritis according to ASAS criteria
* Being able to understand and follow the exercise commands
* Willingness to participate in the study

Exclusion Criteria:

* Trauma history related to cervical region
* A completed ankylosis in cervical region
* Surgery history related to cervical region
* Any vestibular disorders
* Upper extremity involvement other than axial spondyloarthritis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Cervical Proprioception Accuracy | At baseline and six weeks later
  Cervical position error method was used to determine the cervical proprioception accuracy. Cervical position error was evaluated in flexion, extension, rotation and lateral flexion directions and was calculated using a special formula. The results were analyzed as angles.

CONTACTS AND LOCATIONS:
Overall Officials: Deniz Bayraktar, PT, PhD, Principal Investigator — Izmir Katip Celebi University
Locations (1):
- Izmir Katip Celebi University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Data will be sent upon a reasonable request.
Time Frame: December 2022 to December 2042
Access Criteria: Data will be sent for academical purposes (for conducting a meta-analysis or systematic review)

REFERENCES:
- [Background] Sieper J, Braun J, Dougados M, Baeten D. Axial spondyloarthritis. Nat Rev Dis Primers. 2015 Jul 9;1:15013. doi: 10.1038/nrdp.2015.13. PMID 27188328
- [Background] Swinkels A, Dolan P. Spinal position sense and disease progression in ankylosing spondylitis: a longitudinal study. Spine (Phila Pa 1976). 2004 Jun 1;29(11):1240-5. doi: 10.1097/00007632-200406010-00014. PMID 15167664
- [Background] Roijezon U, Clark NC, Treleaven J. Proprioception in musculoskeletal rehabilitation. Part 1: Basic science and principles of assessment and clinical interventions. Man Ther. 2015 Jun;20(3):368-77. doi: 10.1016/j.math.2015.01.008. Epub 2015 Jan 29. PMID 25703454
- [Background] Armstrong B, McNair P, Taylor D. Head and neck position sense. Sports Med. 2008;38(2):101-17. doi: 10.2165/00007256-200838020-00002. PMID 18201114
- [Background] Treleaven J. Sensorimotor disturbances in neck disorders affecting postural stability, head and eye movement control--Part 2: case studies. Man Ther. 2008 Jun;13(3):266-75. doi: 10.1016/j.math.2007.11.002. Epub 2008 Jan 3. PMID 18180194
- [Background] Alahmari K, Reddy RS, Silvian P, Ahmad I, Nagaraj V, Mahtab M. Intra- and inter-rater reliability of neutral head position and target head position tests in patients with and without neck pain. Braz J Phys Ther. 2017 Jul-Aug;21(4):259-267. doi: 10.1016/j.bjpt.2017.05.003. Epub 2017 May 19. PMID 28558952
- [Background] Jull G, Falla D, Treleaven J, Hodges P, Vicenzino B. Retraining cervical joint position sense: the effect of two exercise regimes. J Orthop Res. 2007 Mar;25(3):404-12. doi: 10.1002/jor.20220. PMID 17143898